CLINICAL TRIAL: NCT03739632
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled Study to Explore the Effective Doses and to Assess the Safety and Efficacy of Hypidone Hydrochloride Tablets in Patients With Major Depressive Disorder
Brief Title: Study to Explore the Effective Doses and to Assess the Safety and Efficacy of Hypidone Hydrochloride Tablets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Huahai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYP202-CTP
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 10 mg of Hypidone Hydrochloride tablets (Experimental): Hypidone Hydrochloride tablets 10mg/day Study,5mg tablet is to be given orally, twice daily, for 6 weeks
  Interventions: Drug: Hypidone Hydrochloride tablets
- 20 mg of Hypidone Hydrochloride tablets (Experimental): Hypidone Hydrochloride tablets 20mg/day Study,10mg tablet is to be given orally, twice daily, for 6 weeks
  Interventions: Drug: Hypidone Hydrochloride tablets
- 40 mg of Hypidone Hydrochloride tablets (Experimental): Hypidone Hydrochloride tablets 40mg/day Study,20mg tablet is to be given orally, twice daily, for 6 weeks
  Interventions: Drug: Hypidone Hydrochloride tablets
- comparator (Placebo Comparator): Placebo tablets is to be given orally, twice daily, for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hypidone Hydrochloride tablets — Hypidone Hydrochloride tablets will be given orally, twice daily, for 6 weeks
  Arms: 10 mg of Hypidone Hydrochloride tablets; 20 mg of Hypidone Hydrochloride tablets; 40 mg of Hypidone Hydrochloride tablets
Other: Placebo — Placebo tablets will be given orally, twice daily, for 6 weeks
  Arms: comparator

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Hypidone Hydrochloride tablets in treatment of patients with major depressive disorder (MDD) by evaluating the change of MADRS total scores from baseline to week 6.

DETAILED DESCRIPTION:
A total of 240 major depressive disorder (MDD) subjects between the ages of 18-65 who have current major depressive disorder diagnosed by DSM-5 will be recruited, Eligible patients will be randomized with a 1:1:1:1 ratio into the 4 treatment arms to receive either Hypidone Hydrochloride tablets or placebo, and will be accepted into the protocol after review and providing voluntary written informed consent forms and completion of a comprehensive medical and psychiatric history, physical examination, mental status examination, and routine laboratory assessment.

The subjects will accept the drug treatment twice daily orally for 6 weeks. During the treatment follow up will occur at 8±1 days after treatment, 15±1 days after treatment, 29±2 days after treatment , 43±2 days after treatment to evaluate the safety and efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient or Inpatient, 18-65 years old, male or female
2. Current major depressive disorder diagnosed by DSM-5, single episode(296.21, 296.22, 296.23), or recurrent episode(296.31, 296.32, 296.33)
3. Montgomery-Åsberg Depression Rating Scale (MADRS) total scores in both Screening and Baseline ≥ 26
4. The first item of MADRS in both Screening and Baseline ≥ 3
5. CGI-S in both Screening and Baseline ≥ 4
6. Able to provide written informed consent forms

Exclusion Criteria:

1. Subjects accord with other mental disorders diagnosed by DSM-5
2. Subjects who attempted to suicide, or who presently have a high risk of suicide, or with the tenth item (Suicidal ideation) of C-SSRS ≥ 3
3. Baseline total scores compared with the screening period, the reduction rate of MADRS ≥ 25%
4. Subjects with serious or uncontrolled cardiovascular disease, liver disease, kidney disease, blood disease, endocrine disease, respiratory disease
5. Subjects with clinically significant ECG abnormal (Male QTcF ≥ 450 msec, Female QTcF ≥ 470 msec)
6. Treatment with a MAOI within the 2 weeks prior to the first dose of trial medication
7. Practicing 2 different treatment methods of antidepressants as recommended dose of full course (≥6 weeks)
8. Subjects who have had a Vagus Nerve Stimulation (VNS) device implanted, or who have received Modified Electric Convulsive Therapy (MECT) or Transcranial Magnetic Stimulation (TMS) within 3 months of Screening, or who received light treatment, laser treatment, acupuncture and other Chinese medicine treatment, biofeedback treatment within 2 weeks of Screening
9. Subjects with a history of true allergic response to more than 1 class of medications
10. Subjects who participated in a clinical trial within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline,43 days after treatment
  Change from baseline in MADRS scores，the *total* score ranges[0,60],higher values represent a worse outcome

SECONDARY OUTCOMES:
Hamilton Depression Scale 17 items(HAMD17) | Baseline,43 days after treatment
  Change from baseline in HAMD17 scores,the *total* score ranges[0,50],higher values represent a worse outcome
Hamilton Anxiety Rating Scale (HAM-A) | Baseline,43 days after treatment
  Change from baseline in HAM-A scores,the *total* score ranges[0,56],higher values represent a worse outcome
Clinical Global Impression of Severity Scale(CGI-S) | Screening,Baseline, 8 day after treatment,15 day after treatment,29 day after treatment,43 day after treatment
  Change from baseline in CGI-S scores,the *total* score ranges[0,7],higher values represent a worse outcome
Clinical Global Impression of Improvement Scale(CGI-I) | 8 day after treatment,15 day after treatment,29 day after treatment,43 day after treatment
  the *total* score ranges[0,7],higher values represent a worse outcome
Change in Digit Symbol Substitution Test (DSST) | Baseline, 43 days after treatment
Change in Trail Making Test Parts A&B (TMT) | Baseline, 43 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (19):
- China (19):
  - Beijing Anding Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Guangzhou Hui'ai Hospital, Guangzhou, Guangdong
  - Hebei Mental Health Center, Baoding, Hebei
  - Henan Psychiatric Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Jiangxi Mental Hospital, Nanchang, Jiangxi
  - Jilin Neuropsychiatric Hospital, Siping, Jilin
  - Shandong Mental Health Center, Jinan, Shandong
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Xi'an Mental Health Center, Xi’an, Shanxi
  - The 7th People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - the First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - The Third People's Hospital of Huzhou, Huzhou, Zhejiang
  - Ningbo Kangning Hospital, Ningbo, Zhejiang